CLINICAL TRIAL: NCT05491538
Title: Acceptability and Feasibility of Work-Oriented, Veteran-Centric, Social-Cognitive Skills Training
Brief Title: Acceptability and Feasibility of Work-Oriented Social-Cognitive Skills Training for Veterans With Serious Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4068-P
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Stress Disorder, Post-Traumatic
Keywords: social cognition; employment, supported; psychotherapy, group; mental health
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a single-group, open pilot trial in which participants will receive a group-based social-cognitive skills training program in addition to supported employment services.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Social Cognition and Interaction Training-Work Edition (Experimental): Social Cognition and Interaction Training-Work Edition is a group-based, skills training group that will be offered to participants after they enroll in supported employment.
  Interventions: Behavioral: Social Cognition and Interaction Training-Work Edition (SCIT-WE)

INTERVENTIONS:
Behavioral: Social Cognition and Interaction Training-Work Edition (SCIT-WE) — Participants will attend 1 2-hour skills training group weekly for 13 weeks after enrolling in supported employment. In addition to the group session, participants have a 15-30 minute individual session with the group facilitator weekly to review homework and complete a 10-15 minute exercise with their employment specialist each week to practice skills outside of group. The 13-week skills group is followed by 10 skills review/application sessions conducted during 10 supported employment sessions in the next 13 weeks.

SUMMARY:
Many individuals with serious mental illness have difficulty accurately interpreting interpersonal cues and effectively engaging in social exchanges. Difficulties related to the interpersonal aspects of work can lead to isolation, poor productivity, and job loss. The goals of this study are to: 1) adapt an evidence-based social cognitive skills intervention for work settings and use with Veterans, 2) examine the acceptability of the work focused skills training intervention, 3) assess the feasibility of combining the social cognitive skills training program with supported employment, and 4) examine change on functional outcomes.

The current study will use feedback from veteran and employment specialist stakeholders to adapt an evidence-based social cognitive skills training program, Social Cognition and Interaction Training (SCIT). The intervention will be modified to tailor it to work relationships and to address any unique relationship concerns among Veterans that are identified by stakeholders. SCIT-Work Edition (SCIT-WE) will add: 1) education about work-related social norms; 2) examples of work-related social interactions that require perspective taking and problem- solving; 3) individual sessions with the study therapist to enhance learning and relevance to each participant's goals; 4) structured interactions with the participant's employment specialist to practice skills outside of group; and 5) skill application sessions with the participant's employment specialist that prompt use of skills after training is completed.

SCIT-WE will be developed and piloted in an open trial with 20 Veterans enrolled in the supported employment program at the Minneapolis VA who have a qualifying serious mental illness diagnosis. SCIT-WE will be offered for 2 hours weekly over 13 weeks, when most participants are in the job development and job search phases of supported employment. While participating in the group skills training, participants will have weekly, individual homework review sessions with the group facilitator to promote understanding of the skills and to discuss relevance of the skills to personal goals. Participants also will practice skills weekly with their employment specialist for 10-15 minutes to promote use of skills outside of group sessions. In the 3-months following skills training completion, participants will complete 10 15-minute skills review sessions with their employment specialist to encourage continued skill application in a work setting.

Participants will complete assessments at baseline, before receiving the intervention; 3-months post-enrollment, after participating in a weekly skills training group; and 6-months post-enrollment, after receiving 10 additional individual skills review sessions with their employment specialist. Accessibility will be measured with rate of treatment uptake, rate of treatment completion, and participant attitudes toward the intervention. Feasibility of the intervention will be assessed by examining retention in supported employment and the study at 3- and 6-months post-enrollment. Impact of the intervention will be examined with measures of quality of life, social adjustment, self-efficacy, and work relationship quality. It is hypothesized that the intervention will be acceptable to Veterans. The investigators predict a 50% treatment uptake rate, a 70% intervention completion rate, and positive ratings on measures of satisfaction, interest, and value. The investigators hypothesize that it will be feasible to complete this intervention in combination with supported employment activities. The investigators predict that retention in both skills training and supported employment will be 75% at 3-months post-enrollment and 60% 6-months post enrollment. The investigators hypothesize that positive change will be seen at 3-months post-enrollment and sustained at 6-months post-enrollment on measures of quality of life and social adjustment. The investigators predicted that self-efficacy regarding return to work will be improved at 3-months post-enrollment. The investigators predict that Veterans will report being productive and having positive work relationships 6-months post-enrollment.

The findings will inform the development of a novel intervention targeting the social and functional impairments associated with serious mental illness. The knowledge gained from this study will guide the development of the next generation of interventions. Given that employment is a critical part of recovery, advancement in therapeutic interventions that support Veterans in this process will be of significance.

DETAILED DESCRIPTION:
Rationale and Study Aims: Many individuals with serious mental illness have difficulty accurately interpreting interpersonal cues and effectively engaging in social exchanges. Difficulties related to the interpersonal aspects of work can lead to isolation, poor productivity, and job loss. As a contributor to role functioning, social cognitive ability has become an intervention target. The most established intervention, Social Cognition and Interaction Training (SCIT), is a group psychotherapy that targets 3 social cognitive domains: emotion recognition, theory of mind, and attributional bias. SCIT offers 20-24 hours of instruction and has been delivered to individuals with schizophrenia, bipolar disorder, and depression previously. The goals of this study are to: 1) adapt SCIT for work settings and use with Veterans, 2) examine the acceptability of the work focused skills training intervention, 3) assess the feasibility of combining the social cognitive skills training program with supported employment, and 4) examine change on functional outcomes.

Intervention Development: The SCIT curriculum has three phases. Phase 1 focuses on the role of emotions in social situations and recognizing emotion in self and others. Phase 2 focuses on increasing awareness of cognitive biases and teaching strategies to avoid jumping to conclusions. Phase 3 focuses on integrating skills and applying them to social situations through a social problem-solving process. Social Cognition and Interaction Training-Work Edition (SCIT-WE) will follow the same three phase structure as SCIT. Based upon feedback from stakeholders, this curriculum will be expanded. To contextualize the intervention for work settings and for use with a Veteran population, semi-structured stakeholder interviews will be conducted with Veterans who have participated in supported employment in the previous five years (n = 20) and employment specialists at the Minneapolis VAHCS (n = 5). Stakeholders will be asked about work experiences, work-related social problems that are commonly encountered/observed, types of training/feedback currently received through the supported employment program, feedback about additions to the curriculum, and concerns about the proposed integration of SCIT-WE with supported employment. Notes will be taken during the interviews and used to identify educational topics and types of skills training that would be most useful additions to the curriculum.

Four to six hours of content will be added to the SCIT group session curriculum focused on workplace social norms, expression and regulation of emotion at work, and communication styles. In addition, training materials will be developed to supplement the SCIT curriculum: (1) standardized homework assignments that reinforce the SCIT curriculum with work-related scenarios; (2) standardized activities that participants can complete with their employment specialist to practice skills outside of sessions; (3) standardized skill application session materials to prompt continued use of skills after training sessions are completed; and (4) materials to standardize communications between the study therapist and the employment specialists.

An open trial pilot study will be conducted with 20 Veterans who are outpatients and enrolled to receive supported employment services at the Minneapolis VA Health Care System. Veterans participating in supported employment are receiving services from a mental health team, are motivated to pursue employment, and are seeking employment within 30 miles of the medical center. Veterans will be provided with information about the study after enrollment in supported employment. Veterans who express an interest in the study will complete a screening interview that establishes psychiatric diagnosis and eligibility for the study.

Veterans who choose to enroll in the study will attend one 2-hour SCIT-WE session weekly for 13 weeks, when most participants are in the job development and job search phases of supported employment. Group size will be 4 or fewer Veterans. The group will be facilitated by a doctoral level therapist who has received training from one of the intervention developers and who has over five years of experience offering SCIT to Veterans. To promote generalization of skills training, weekly homework and practice partner assignments will be given to participants to complete outside of group. The group facilitator will contact participants by phone each week for a 15-30-minute individual review of assigned homework and to discuss its relevance to their personal goals. Veterans will complete the practice partner assignments during sessions with their employment specialist. Practice partner activities will take 10-15 minutes to complete in session. These activities are an opportunity for the Veteran to practice using a skill introduced during group with someone outside of group. While a Veteran is participating in SCIT-WE, the group facilitator will contact the employment specialist at the end of each training phase to provide feedback about the Veteran's social cognitive performance. Upon completion of SCIT-WE skills training group, Veterans will continue to meet with their employment specialist for supported employment activities. In the 3 months post-skills training, employment specialists will use structured intervention materials developed for SCIT-WE during 10 sessions to prompt skill application. This material will add 15 minutes to their sessions with participants.

Assessments: To evaluate the intervention, participants will complete assessments at baseline, before receiving the intervention; 3-months post-enrollment, after participating in a weekly skills training group; and 6-months post-enrollment, after receiving 10 additional individual skills review sessions with their employment specialist. Accessibility will be measured with rate of treatment uptake, rate of treatment completion, and participant attitudes toward the intervention. Feasibility of the intervention will be assessed by examining retention in supported employment and the study at 3- and 6-months post-enrollment. Impact of the intervention will be examined with measures of quality of life, social adjustment, self-efficacy, and work relationship quality. It is hypothesized that the intervention will be acceptable to Veterans. The investigators predict a 50% treatment uptake rate, a 70% intervention completion rate, and positive ratings on measures of satisfaction, interest, and value. The investigators hypothesize that it will be feasible to complete this intervention in combination with supported employment activities. The investigators predict that retention in both skills training and supported employment will be 75% at 3-months post-enrollment and 60% 6-months post enrollment. The investigators hypothesize that positive change will be seen at 3-months post-enrollment and sustained at 6-months post-enrollment on measures of quality of life and social adjustment. The investigators predicted that self-efficacy regarding return to work will be improved at 3-months post-enrollment. Direction and magnitude of change will be measured with Cohen's d and 95% confidence intervals. The investigators predict that veterans will report being productive and having positive work relationships 6-months post-enrollment.

Treatment Manual Development: To gain additional insights about the experience of the intervention for participants, an exit interview will be completed 6-months post-enrollment. Veterans who enroll in the open trial pilot (n = 20) and employment specialists (n = 5) who use the educational materials developed for this project will each complete a 90-minute, semi-structured exit interview. The interview will assess: (1) attitudes about the intervention components, structure, and materials; (2) suggestions for intervention improvement; (3) impact of the training on intervention targets and unexpected impacts; and (4) barriers and facilitators to training participation. Interviews will be conducted by phone or in-person by a doctoral level clinician. Exit interviews will be transcribed and processed using an efficient, rapid turn-around analytic approach to identify key themes. Based upon participant feedback, a SCIT-WE treatment manual will be finalized for use in future research.

Significance: The findings will inform the development of a novel intervention targeting the social and functional impairments associated with serious mental illness. The knowledge gained from this study will guide the development of the next generation of interventions. Given that employment is a critical part of recovery, advancement in therapeutic interventions that support Veterans in this process will be of significance.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who are outpatients and enrolled to receive supported services at the Minneapolis VA Health Care System.
* Veterans are eligible for this program if they are receiving services from a mental health team at the Minneapolis VA Health Care System, are motivated to pursue employment, and are seeking employment within 30 miles of the medical center.
* Veterans will be eligible for the study if they have a DSM-5 diagnosis of Schizophrenia, Schizoaffective Disorder, Bipolar I Disorder, Bipolar II Disorder, Recurrent Major Depressive Disorder, or PTSD.

Exclusion Criteria:

Study exclusion criteria are:

* presence of a moderate or severe traumatic brain injury
* presence of a cognitively compromising neurological disease
* understanding of English that is not sufficient for comprehension of testing procedures
* premorbid IQ less than 70
* behavior that prevents participation in a group intervention
* hearing or visual impairment that prevents completion of intervention and testing procedures
* clinical instability, defined as active suicidal ideation or hospitalization in the previous 4 weeks
* current diagnosis of alcohol or substance use disorder, severe
* current participation in another mental health intervention study
* inability to commit to 7-9 months of study participation due to a planned move or unstable housing
* inability to provide informed consent
* presence of a guardian of person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-11-27 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Social Adjustment Scale-Self-Report: Short Version (SAS-SR: Short) Change | Baseline and 3 months
  This task is a 24-item self-report scale that assesses functioning in 6 social roles in the prior 2 weeks. Total score is a T-score and ranges from 0-100. A higher score indicates more impairment in social role functioning.
Social Adjustment Scale-Self-Report: Short Version (SAS-SR: Short) Change | Baseline and 6 months
  This task is a 24-item self-report scale that assesses functioning in 6 social roles in the prior 2 weeks. Total score is a T-score and ranges from 0-100. A higher score indicates more impairment in social role functioning.
Recovering Quality of Life (ReQoL)-20 Change | Baseline and 3 months
  This task is a 20-item self-report, recovery-focused quality of life measure. Total score ranges from 0-80. A higher score indicates greater quality of life.
Recovering Quality of Life (ReQoL)-20 Change | Baseline and 6 months
  This task is a 20-item self-report, recovery-focused quality of life measure. Total score ranges from 0-80. A higher score indicates greater quality of life.
Return to Work Self-Efficacy Scale (RTW-SE) Change | Baseline and 3 months
  This 11-item self-report scale measures self perception of ability to return to work the next day. Total score ranges from 11 to 66. A higher score indicates greater self-confidence in ability to work.
Intrinsic Motivation Inventory - Interest subscale | 3 months
  This subscale measures self-report of interest and enjoyment from an activity on a 7-point scale. Total score ranges from 1-7, with a higher score indicating greater interest in the training activity. The 3-month measurement will reflect interest and enjoyment in the skills training group.
Intrinsic Motivation Inventory - Interest subscale | 6 months
  This subscale measures self-report of interest and enjoyment from an activity on a 7-point scale. Total score ranges from 1-7, with a higher score indicating greater interest in the training activity. The 6-month measurement will reflect interest and enjoyment in the individual skills review sessions.
Intrinsic Motivation Inventory - Value subscale | 3 months
  This subscale measures self-report of perceive value and importance of an activity on a 7-point scale. Total score ranges from 1-7, with a higher score indicating greater value in the training activity. The 3-month measurement will reflect value and importance of the skills training group.
Intrinsic Motivation Inventory - Value subscale | 6 months
  This subscale measures self-report of perceive value and importance of an activity on a 7-point scale. Total score ranges from 1-7, with a higher score indicating greater value in the training activity. The 6-month measurement will reflect value and importance of the individual skills review sessions.
Client Satisfaction Questionnaire (CSQ-8) | 3 months
  This questionnaire is an 8-item self-report measure of satisfaction with health services. Total score ranges from 8-32. A higher score indicates greater satisfaction with services. The 3-month measurement will reflect satisfaction with the skills training group.
Client Satisfaction Questionnaire (CSQ-8) | 6 months
  This questionnaire is an 8-item self-report measure of satisfaction with health services. Total score ranges from 8-32. A higher score indicates greater satisfaction with services. The 6-month measurement will reflect satisfaction with the individual skills review sessions.
Rate of Treatment Uptake | Recruitment
  Percentage of eligible participants who express interest in the intervention
Completer of Skills Training Intervention | 3 months
  Percentage of sample that qualifies as completing the intervention. A participant is defined as a completer is they attend 80% or more of intervention sessions.
Retention in supported employment | 3 months
  Percentage of study participants who remain involved in supported employment 3 months post-enrollment.
Retention in supported employment | 6 months
  Percentage of study participants who remain involved in supported employment 6 months post-enrollment.
Retention in skills training program | 3 months
  Percentage of study participants who remain enrolled in the study 3 months post-enrollment.
Retention in skills training program | 6 months
  Percentage of study participants who remain enrolled in the study 6 months post-enrollment.

SECONDARY OUTCOMES:
Mentoring and Communication Support Scale (MCSS) | 6 months
  This scale is a self-report measure of perceived relationship quality with colleagues and supervisors at work. The scale has four subscales: Collegial Support, Task Support, Career Mentoring, and Coaching. Collegial Support and Task Support scales indicate the amount of support perceived from co-workers, emotionally and in terms of conveying knowledge about how to do the job. The scales range from 4-20 with a higher score indicating a greater level of perceived support. Career Mentoring and Coaching scales measure support perceived from supervisor in terms of advice as well as instruction on how to do one's job. The Career Mentoring scale ranges from 4-20, with a higher score indicating more support. The Coaching scale ranges from 3-15, with a higher score indicating more support.
Vocational Efficacy in Trauma Survivors Scale | 6 months
  This scale is a self-report measure of perceived social support and efficacy coping with mental health symptoms at work. The scale has two subscales: Self Disclosure and Workplace Coping. The Self Disclosure subscale ranges from 4-20, with a higher score indicating greater comfort self disclosing about mental health issues at work. The Workplace Coping subscale ranges from 7-35, with a higher score indicating greater confidence in one's abilities to manage mental health symptoms at work.
Work Limitations Questionnaire (WLQ) | 6 months
  This measure is a self-report scale that provides work performance information in four domains: Mental-Interpersonal, Time Management, Output, and Physical Demands. The At-Work Productivity Loss Summary score reflects the percentage of time that the individual had job performance deficits due to mental or physical health problems in the prior 2 weeks. A higher score indicates poorer performance.

CONTACTS AND LOCATIONS:
Overall Officials: Tasha Marie Nienow, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
There is plan to make individual participant data sets available to others. Final, de-identified final datasets that underlie publications will be made available upon written request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Final datasets will be available at study completion in November 2024. They will remain available for at least 6 years post study closure.
Access Criteria: De-identified data will be made available so that analyses can be re-run, secondary analyses can be completed, and study data can be included in future meta-analyses. When the principal investigator receives a request from another investigator, the dataset and the request will be reviewed by the principal investigator and Minneapolis VA Privacy Officer prior to release.